CLINICAL TRIAL: NCT00150540
Title: A Long Term, Open Label Extension Study of Protocols LAM-IV-301, LAM-IV 303, LAM-IV 307 AND LAM-IV 308.
Brief Title: A Long Term Study of Lanthanum Carbonate in Patients Requiring Dialysis Who Have Ived Lanthanum Carbonate in Previous Studies Defined by the Protocol.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-309
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate

SUMMARY:
The purpose of this study is to assess the safety of lanthanum carbonate in patients undergoing dialysis who have received lanthanum carbonate in the previous studies and wish to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in LAM-IV-301, LAM-IV-303, LAM-IV-307 OR LAM-IV-308 and received lanthanum carbonate
* Patients must continue to require treatment with a phosphate binder for hyperphosphatemia
* male or non-pregnant female who agrees to use an effective contraceptive method while on study treatment and for 30 days thereafter

Exclusion Criteria:

* Patients withdrawn from LAM-IV-301, LAM-IV-303 OR LAM-IV-307 prior to randomization
* Patients withdrawn from LAM-IV-301, LAM-IV-303, LAM-IV-307 OR LAM-IV-308 due to adverse events termed "possible" or "related" to study medication
* Pregnant or lactating women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93
Dates: Start 2002-10-14 (Actual); Primary Completion 2005-06-29 (Actual); Study Completion 2005-06-29 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Up to 24 months

SECONDARY OUTCOMES:
Changes in pre-dialysis serum phosphate levels | Baseline, Months 3, 6, 9, 12, 15, 18, 21, 24.
Control of pre-dialysis serum phosphate levels | Baseline, Months 3, 6, 9, 12, 15, 18, 21, 24.
Plasma lanthanum levels | Baseline, Months 3, 6, 9, 12, 15, 18, 21, 24.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda